CLINICAL TRIAL: NCT02040220
Title: Special Drug Use Investigation of EYLEA for CRVO
Brief Title: Prospective, Non-interventional, Multi-center Post-authorization Safety Study of Eylea for Central Retinal Vein Occlusion (CRVO)
Acronym: JPMS-CRVO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 16641; EYL-CRVO (Other: company internal)
Record Dates: First submitted 2014-01-08; First posted 2014-01-20 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Retinal Vein Occlusion
Keywords: CRVO, Macular edema, Aflibercept, anti-VEGF
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Eylea treatment goup
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — 2 mg of Eylea will be treated per one injection at more than one months interval usually.

SUMMARY:
This is a prospective, non-interventional, multi center post-authorization safety study that includes patients with a diagnosis of CRVO. The investigator will have made the choice of treatment (EYLEA) as well as the decision to use EYLEA according the Japanese Package Insert prior to enrolling the patient in this study.

The observation period for each patient starts when therapy with EYLEA is initiated. The enrollment period is 2 years. Patients will be followed for a time period of 2 years or until it is no longer possible (e.g. lost to follow-up) within the 2 years.

For each patient, data are collected as defined in the case report form at the initial visit, follow-up visits and final visit, either by routine clinical visits (as per investigators routine practice).

There will interim analysis of study data: 6 months after last patient first visit and J-PSUR(Japanese-Periodic Safety Update Report )

ELIGIBILITY:
Inclusion Criteria:

* Patients who start EYLEA treatment for CRVO

Exclusion Criteria:

* Patients who have already received EYLEA treatment
* Patients who are contraindicated based on approved label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients with a diagnosis of CRVO will be enrolled after the decision for treatment with EYLEA has been made by the investigator. Those patients prescribed EYLEA previously will not be included in this study. Physicians should consult the full prescribing information for EYLEA before enrolling patients and familiarize themselves with the safety information in the product package label. Eligible patients who receive EYLEA will be enrolled and documented in the eCRF.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Number of episodes of adverse drug reactions and adverse events(serious or non-serious, related or not related, ocular or non ocular) | 6 months after start of treatment with the drug

SECONDARY OUTCOMES:
Effectiveness (visual acuity) | 6months after start of treatment with the drug
Effectiveness (retina thickness) | 6months after start of treatment with the drug

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan